CLINICAL TRIAL: NCT03273075
Title: Pharmacokinetic/Pharmacodynamic Effects of add-on Antiplatelet Therapy With Parenteral Cangrelor as Compared to Standard Dual Antiplatelet Treatment in Patients With ST-elevation Myocardial Infarction Complicated by Out-of-hospital Cardiac Arrest and Treated With Targeted Temperature Management
Brief Title: Add-on Cangrelor in STEMI-triggered Cardiac Arrest
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alexander Spiel, Assoc.Prof. Priv.Doz. Dr.med.univ. Alexander Spiel, Medical University of Vienna
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cang 2016-003265-26
Record Dates: First submitted 2017-08-23; First posted 2017-09-06 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Cardiopulmonary Arrest With Successful Resuscitation; ACS - Acute Coronary Syndrome; Hypothermia, Induced
Keywords: P2Y12r inhibitor; Cardiac Arrest; STEMI; HTPR
MeSH Terms: conditions — Acute Coronary Syndrome; Hypothermia; Heart Arrest; ST Elevation Myocardial Infarction | interventions — cangrelor; Saline Solution; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Prasugrel + Cangrelor (Active Comparator): If eligible, assigned to this arm and without contraindications to prasugrel administration, patients will receive a loading dose of prasugrel (60 mg) via nasogastric tube as soon as possible after arrival at the emergency department. Afterwards a 30 micrograms (mcg)/kg iv bolus of cangrelor followed immediately by a 4 mcg/kg/min iv infusion (lasting for at least 2 hours or for the duration of the revascularization procedure, whichever is longer) will be administered.
  Interventions: Drug: Cangrelor; Drug: Prasugrel
- Ticagrelor + Cangrelor (Active Comparator): If eligible and assigned to this arm (i.e. patients who have contraindications against prasugrel (age >75years, weight <60kg, history of transient ischemic attack, ischemic stroke, intracranial bleeding, known allergy against prasugrel/Efient), patients will receive a loading dose of ticagrelor (180 mg) via nasogastric tube as soon as possible after arrival at the emergency department. Afterwards a 30 micrograms (mcg)/kg iv bolus of cangrelor followed immediately by a 4 mcg/kg/min iv infusion (lasting for at least 2 hours or for the duration of the revascularization procedure, whichever is longer) will be administered.
  Interventions: Drug: Cangrelor; Drug: Ticagrelor
- Prasugrel + Placebo (Placebo Comparator): If eligible, assigned to this arm and no contraindications to prasugrel, patients will receive a loading dose of prasugrel (60 mg) via nasogastric tube as soon as possible after arrival at the emergency department.
  Afterwards a 30 micrograms (mcg)/kg iv bolus of placebo (0.9% NaCl) followed immediately by a 4 mcg/kg/min iv infusion of placebo (0.9% NaCl) (lasting for at least 2 hours or for the duration of the revascularization procedure, whichever is longer) will be administered.
  Interventions: Drug: Placebo; Drug: Prasugrel
- Ticagrelor + Placebo (Placebo Comparator): If eligible and assigned to this arm (i.e. patients who have contraindications against prasugrel (age >75years, weight <60kg, history of transient ischemic attack, ischemic stroke, intracranial bleeding, known allergy against prasugrel/Efient), patients will receive a loading dose of ticagrelor (180 mg) via nasogastric tube as soon as possible after arrival at the emergency department.
  Afterwards a 30 micrograms (mcg)/kg iv bolus of placebo (0.9% NaCl) followed immediately by a 4 mcg/kg/min iv infusion placebo (0.9% NaCl) (lasting for at least 2 hours or for the duration of the revascularization procedure, whichever is longer) will be administered.
  Interventions: Drug: Placebo; Drug: Ticagrelor

INTERVENTIONS:
Drug: Cangrelor — The intervention comprises add-on Cangrelor infusion (administration in compliance with manufacturer instructions) in addition to and after administration of standard P2Y12-blocker (prasugrel or ticagrelor) therapy.
  Arms: Prasugrel + Cangrelor; Ticagrelor + Cangrelor
Drug: Placebo — The intervention comprises add-on placebo infusion (0.9% NaCl) in addition to and after administration of standard P2Y12-blocker (prasugrel or ticagrelor) therapy as placebo comparator
  Other Names: 0.9% NaCl
  Arms: Prasugrel + Placebo; Ticagrelor + Placebo
Drug: Prasugrel — The intervention comprises the standard P2Y12-blocker prasugrel therapy if not contraindicated.
  Arms: Prasugrel + Cangrelor; Prasugrel + Placebo
Drug: Ticagrelor — The intervention comprises the standard P2Y12-blocker ticagrelor therapy if prasugrel is contraindicated and no contraindication to ticagrelor is present.
  Arms: Ticagrelor + Cangrelor; Ticagrelor + Placebo

SUMMARY:
In patients with ST-elevation myocardial infarction (STEMI) undergoing percutaneous coronary angioplasty (PCI) P2Y12 receptor (P2Y12r) inhibition should be achieved as soon as possible. Resuscitated STEMI-patients receiving targeted temperature management (TTM, therapeutic hypothermia) after cardiac arrest, however, show deteriorated and delayed early response to available oral P2Y12r inhibitors. Therapeutic hypothermia attenuates the drugs' effectiveness by reducing its gastrointestinal absorption and metabolic activation. Acute stent thrombosis is 5-fold increased after angioplasty following resuscitated cardiac arrest because of insufficient early platelet suppression. Thus, aggressive antiplatelet strategies are needed to achieve optimal platelet suppression during PCI in those patients. The first intravenous P2Y12r inhibitor, cangrelor, has recently received marketing authorization for the acute treatment of STEMI. We hypothesize that add-on antiplatelet therapy with intravenous Cangrelor on-top of standard dual anti platelet therapy (DAPT) with Prasugrel or Ticagrelor is superior to standard antiplatelet therapy alone in terms of suppressing ADP-dependent platelet activation in resuscitated STEMI-patients receiving TTM.

DETAILED DESCRIPTION:
Neurologic damage after cardiac arrest is frequent and therapeutic options to improve neurological outcome are limited. Treatment by therapeutic hypothermia (TH, 32-34◦C) for 12-24 h showed improved neurological outcome in several trials. Therefore, international guidelines recommend targeted temperature management (TTM) to 32-34◦C (or at least 36°C) for 12-24 h, especially when the initial rhythm was ventricular fibrillation.

However, patients treated with TTM after cardiac arrest show deteriorated and delayed response to P2Y12 receptor (P2Y12r) inhibitors as determined by platelet reactivity index vasodilator-stimulated phosphoprotein phosphorylation (PRI VASP) after administration of the loading dose of clopidogrel, prasugrel and ticagrelor. Especially the response to clopidogrel is poor with up to >80% non-responder after 24 hours. Impaired P2Y12r blockade may lead to acute stent-thrombosis and trigger overall adverse outcome.

There are several explanations for the impaired efficacy of P2Y12r inhibitors in cardiac arrest patients. First, marketed oral P2Y12r inhibitors have to be applied in crushed form via nasogastric tube in comatose post cardiac arrest patients. Placement of nasogastric tube and crushing may delay onset of therapy. Second, drug uptake and bioavailability of oral P2Y12r inhibitors are dependent on gastric motility and sufficient splanchnic blood supply, which is affected by TTM, acute critical illness (shock) and concomitant therapy. Particularly, sedation and analgesic agents, especially concomitant morphine therapy, can hamper gastric emptying. Various recent trials demonstrated that morphine administration delays and attenuates clopidogrel, prasugrel and ticagrelor exposure and action in healthy subjects and patients with myocardial infarction.

The recently authorized parenteral cangrelor is an adenosine triphosphate (ATP) analogue that binds reversibly and with high affinity to the platelet P2Y12r. It induces a highly effective inhibition of ADP-induced platelet aggregation immediately after intravenous (iv) bolus administration and allows for restoration of platelet function within 1-2 h of infusion discontinuation. The pharmacokinetic properties known so far suggest cangrelor being the "ideal" P2Y12r inhibitor for patients with cardiac-ischemia triggered OHCA treated with TH and may overcome the impaired and delayed P2Y12r blockade seen with the oral P2Y12r inhibitors.

Cardiac arrest is a leading cause of death among adults over the age of 40 in the European Union (EU) and other western countries. In the EU alone, more than 400.000 people of all ages experience EMS-assessed out-of-hospital non-traumatic cardiac arrest each year and most of them die. In a large proportion of these patients (about 50%) an acute coronary syndrome (ACS), mainly acute ST-elevation myocardial infarction, leading to ventricular fibrillation and cardiac standstill is the cause of the cardiac arrest. Various trials demonstrated that early cardiac intervention including stent placement to the culprit lesion improves outcome in this patient group. The P2Y12r plays a central role in platelet activation and P2Y12r inhibitors are part of standard care in patients with ACS. Delayed and insufficient P2Y12r inhibition may predispose to acute stent thrombosis with potential devastating effects including cardiogenic shock, re-arrest and death. Given the deteriorated and delayed response to oral P2Y12r inhibitors in cardiac arrest patients treated with TH, clinical evaluation of the recently marketed parenteral P2Y12r inhibitor cangrelor is mandatory in this patient group.

To determine the effect of add-on cangrelor in STEMI-associated out-of-hospital cardiac arrest (OHCA) who receive TTM and are scheduled for PCI, a phase 4 trial will be conducted.The trial consists of 2 parts. Part A (n=12, 8months duration): An open-fashioned pilot safety-study to ensure sufficient platelet suppression (<466AU*min, impedance aggregometry) over 24 hours after concurrent cangrelor-prasugrel/ticagrelor administration. The aim is to determine pharmacokinetics and -dynamics of oral P2Y12r-inhibitors with and without concomitant administration of cangrelor. Part B (n=48, 32months duration): A factorial randomized, placebo-controlled, double-blind study with 4 study cohorts enrolling 48 patients who will first be randomised to receive prasugrel (n=24) or ticagrelor (n=24) and secondly to additionally receive cangrelor or placebo (sterile saline). Primary endpoint: ADP-dependent platelet reactivity at time of stent placement (AU*min). Student's t-test to test H0 (no difference in AU*min, cangrelor vs placebo).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-74 years
* comatose survivors of OHCA
* initial shockable rhythm (i.e. ventricular fibrillation or pulseless ventricular tachycardia)
* STEMI (post-ROSC electrocardiography)
* application of TTM;
* scheduled for PCI
* interval of <10 min from cardiac arrest to initiation of cardiopulmonary
* resuscitation (no-flow interval); interval of <60 min from initiation of cardiopulmonary resuscitation
* to ROSC (low-flow interval)
* eligible for treatment with standard loading doses of DAPT including
* aspirin and either prasugrel or ticagrelor.

Exclusion Criteria:

* Pregnant or breast-feeding patients
* Body weight <60kg
* Response to verbal commands after ROSC
* (thus not eligible for TTM)
* Cardiac arrest due to: trauma, exsanguination, strangulation, smoke
* inhalation, drug overdose, electrocution, hanging or drowning, or intracranial hemorrhage
* Patients not
* achieving ROSC or subjected to an extracorporeal circulatory assist device
* Acute treatment with P2Y12r inhibitor other than prasugrel or ticagrelor
* Active bleeding or increased risk of bleeding because of irreversible coagulation disorders or due to recent major surgery/trauma or uncontrolled
* severe hypertension
* Known history of ischemic or hemorrhagic stroke or transient ischemic attack
* (TIA)
* Known history of severe hepatic impairment (Child Pugh C)
* Known history of severe renal impairment (creatinine clearance <30mL/min)
* Hypersensitivity to the active substance or to any of the excipients
* Terminal illness present before cardiac arrest
* Thrombolysis therapy
* Scheduled for coronary bypass surgery (CABG)
* Prior P2Y12r inhibitor use in the past 7 days
* Prior vitamin K antagonists/NOACs use in past 7 days
* Patients with known allergic reaction to P2Y12r inhibitors.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity at stent placement | up to 4 hours; time from study drug administration (Cangrelor/Placebo) to stent placement
  Platelet reactivity (ADP-dependent platelet inhibition) at the time of cardiac intervention (i.e. at the time of stent placement) measured by impedance aggregometry (Multiplate Analyzer; aggregation units/min, AU*min)

SECONDARY OUTCOMES:
Platelet reactivity | 15 minutes, 30 minutes, 60 minutes, 120 minutes, 240 minutes, 12hours from administration of study drug.
  Platelet reactivity at baseline, 15 minutes, 30 minutes, 60minutes, 120 minutes, 240 minutes and 12 hours after study drug administration (Multiplate Analyzer, AU*min; VASP assay, platelet reactivity units PRU; PFA-100, closure time, CT).
Platelet inhibition | 15 minutes, 30 minutes, 60 minutes, 120 minutes, 240 minutes, 12hours from administration of study drug.
  Onset of ADP-dependent platelet inhibition (Multiplate Analyzer, VASP assay, PFA-100).
Maximum Plasma Concentration [Cmax] | 15 minutes, 30 minutes, 60 minutes, 120 minutes, 240 minutes, 12hours from administration of study drug.
  Prasugrel/Ticagrelor/Cangrelor metabolites will be measured by liquid chromatography-tandem mass spectrometry (LC-MS/MS) at the time of stent placement, 15minutes, 30 minutes, 60 minutes, 120 minutes, 240 minutes and 12 hours after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Alexander o: Spiel, Prof., MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No